CLINICAL TRIAL: NCT00138567
Title: Extension to a Study on the Efficacy and Safety of Vildagliptin Compared to Metformin in Drug Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2309E1
Record Dates: First submitted 2005-08-27; First posted 2005-08-30 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
This is a 52-week extension to a study to assess the safety and effectiveness of vildagliptin, an unapproved drug, compared to metformin in lowering overall blood glucose levels in people with type 2 diabetes who have not been previously treated with drug therapy to lower their blood sugar. The purpose of the extension study is to gather data on the long-term safety and effectiveness of vildagliptin in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Only patients successfully completing study CLAF237A2309 are eligible
* Written informed consent
* Ability to comply with all study requirements

Exclusion Criteria:

* Premature discontinuation from CLAF237A2309
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 78 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 530
Dates: Start 2005-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Safety during 104 weeks of treatment
Change from baseline in HbA1c at 104 weeks

SECONDARY OUTCOMES:
Change in HbA1c between 52 weeks and 104 weeks
Change in fasting plasma glucose between 52 weeks and 104 weeks
Change from baseline in fasting plasma glucose at 104 weeks
Change from baseline in HOMA B at 104 weeks
Change in HOMA B between 52 weeks and 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, East Hanover, New Jersey, United States
- Novartis Investigative site, Investigative Centers, Germany

REFERENCES:
- [Result] Goke B, Hershon K, Kerr D, Calle Pascual A, Schweizer A, Foley J, Shao Q, Dejager S. Efficacy and safety of vildagliptin monotherapy during 2-year treatment of drug-naive patients with type 2 diabetes: comparison with metformin. Horm Metab Res. 2008 Dec;40(12):892-5. doi: 10.1055/s-0028-1082334. Epub 2008 Aug 22. PMID 18726829
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595